CLINICAL TRIAL: NCT06393231
Title: Clinical Study on the End Time of Acupuncture and Moxibustion Therapy for Peripheral Facial Paralysis: Randomized Controlled Trial
Brief Title: Clinical Study on the End Time of Acupuncture and Moxibustion Therapy for Peripheral Facial Paralysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20240123-04-KS-01
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Facial Paralysis
Keywords: peripheral facial paralysis; acupuncture; sequelae
MeSH Terms: conditions — Facial Paralysis | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observation group (Experimental): Sunnybrook score ≥83 points
  Interventions: Other: acupuncture
- control group (Active Comparator): Sunnybrook score ≥95 points
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Acupuncture is applied to ST8, GB14, BL12, SJ23, ST2, SI18, ST4, ST7, RN24, Ex-HN16, SJ17 and LI4 on the affected side and needles are retained for half an hour.Add infrared irradiation therapy in the same time
  Other Names: infrared irradiation therapy; moxibustion

SUMMARY:
Bell's palsy itself has a certain self-healing tendency. Therefore, it is recommended to leave a bit of Bell's palsy for self-recovery without treatment. If complete recovery is achieved after treatment, complications such as stiffness, contracture and even hemifacial inversion may occur as time moves. Therefore, this study aims to evaluate the optimal end time of acupuncture for facial paralysis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, controlled study, with a total of 120 eligible patients randomly divided into an observation group (n=60) and a control group (n=60). Both groups received facial acupuncture combined with infrared irradiation treatment, once a day,10 times as a course, and the next course of treatment will be carried out after a 5-day rest.The treatment duration for both groups will not exceed three months, with the observation group aiming for a Sunnybrook score of ≥83 and the control group aiming for a score≥95. The primary outcome measure is Sunnybrook scores at 6 months after onset compared with baseline. Secondary outcome measures included Sunnybrook Scores, electroneurography, blink reflex, Facial Disability Index, Self-Rating Depression Scale and Self-Rating Anxiety Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75 years.
2. Patients diagnosed with peripheral facial paralysis≤7 days before screening and was the first time.
3. All cases have symptoms and signs or have been examined by CT, MRI, etc., excluding peripheral facial paralysis caused by central nervous system diseases, ear diseases, and trauma.
4. Those who voluntarily sign the Research Informed Consent Form

Exclusion Criteria:

1. Patients with bilateral facial nerve palsy or recurrent facial nerve palsy (more than two occurrences).
2. Pregnant or nursing patients.
3. Patients with critically ill which is difficult to make a definite evaluation of the efficacy and safety of treatment
4. Those who accept other treatment methods or cannot adhere to this plan, which affects the efficacy observation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sunnybrook(SB) score | Change from Baseline scores of SB score at at 6-months after onset.
  This scoring was used to detect the severity of peripheral facial paralysis(PFP).Which include three parts: resting symmetry, symmetry of voluntary movement, and synkinesis. In the resting symmetry scoring of the facial nerve, "normal" in each area refers to being "symmetrical/equivalent" compared to the healthy side. The total score for facial nerve function assessment is calculated as voluntary movement score minus resting symmetry score minus synkinesis score, with a maximum score of 100.The sunnybrook scores were used to define five categories of PFP severity:Normal person（90~100 points）;mild PFP levels（76~89 points）;moderate PFP levels（61~75 points）;moderate to severe PFP levels（31~60points）;and presence of severe PFP（0~30 points）。

SECONDARY OUTCOMES:
Sunnybrook(SB) score | Change from Baseline scores of SB score at at 3、12months after onset.
  This scoring was used to detect the severity of peripheral facial paralysis(PFP).Which include three parts: resting symmetry, symmetry of voluntary movement, and synkinesis. In the resting symmetry scoring of the facial nerve, "normal" in each area refers to being "symmetrical/equivalent" compared to the healthy side. The total score for facial nerve function assessment is calculated as voluntary movement score minus resting symmetry score minus synkinesis score, with a maximum score of 100.The sunnybrook scores were used to define five categories of PFP severity:Normal person（90~100 points）;mild PFP levels（76~89 points）;moderate PFP levels（61~75 points）;moderate to severe PFP levels（31~60points）;and presence of severe PFP（0~30 points）。
Electroneuronography (ENoG) | Change from Baseline amplitude and potential of CAMP and the numbers of pathological ENoG at at 6、12months after onset.
  The goal of the Electroneurography (ENoG) testing is to measure the amount of neural degradation that has occurred distal to the site of facial nerve injury by measuring the muscle response to an electrical stimulus. The testing of ENoG involves recording the compound muscle action potential (CAMP) of the mimetic muscles, including Orbicularis oculi, Frontalis muscle, Orbicularis oris and Zygomaticus muscle. ENoG is performed first on the healthy side of the face and then on the affected side. Nerve damage or nerve fiber degeneration leads to a decrease or loss of the CAMP. The amplitude of the CAMP on the affected side is compared to the CAMP of the healthy side and expressed as percent (amplitude of the paralyzed side divided by the amplitude of the normal side). A side difference of 30% or bigger is considered pathologic.
Blink Reflex | Change from Baseline number of pathological Blink Reflex at 6、12months after onset.
  The blink reflex test is to measures the facial nerve since the blink reflex delivers information on facial nerve function with normal trigeminal function. Blink reflex testing involves electrical stimulation of the supraorbital nerve on the affected side combined with a 2-channel simultaneous surface electromyogram recording from both orbicularis oculi muscles. The exit of the supraorbital nerve in the supraorbital foramen is palpated on the rim of the orbit. Stimulation with 10-20 mA and 0.2 ms duration is used to produce a constant reflex. In blink reflex testing, two responses, R1 and R2, are analyzed. R1 is the fast ipsilateral response of the orbicularis oculi muscle with a latency of about 10-12 ms. The second bilateral response R2 has a latency of about 30-41 ms. The R2 latency differences between both sides higher than 5-8 ms is considered pathologic.
Facial disability index (FDI) | Change from Baseline scores of FDI score at at 3、6、12months after onset.
  The facial disability index (FDI) included the FDI Physical Function Subscale (FDIP) and the FDI Social/Well-being Subscale (FDIS), with a total of 10 questions in each section.The disease severity decreases as the scores rise
Self-Rating Anxiety Scale(SAS) | Change from Baseline scores of FDI score at at 3、6、12months after onset.
  The full name of the scale called Zung Self-Rating Anxiety Scale.The SAS contains 20 questions. Each question is scored on a scale of 1-4 (never, some of the time, relatively often, most of the time). Fifteen questions involve the assessment of increasing anxiety levels, and five questions involve decreasing anxiety levels.Each items points accumulated as raw scores,the lowest raw score is 20 points, the highest raw score is 80 points. The raw scores multiply by 1.25, taking the integer part as the standard scores.The SAS standard scores were used to define four categories of anxiety severity: within normal ranger no significant psychopathology (25-49points);presence of mild to moderate anxiety levels (50-59points); severe anxiety levels (60-69points); and presence of extreme anxiety (70-100points).
Self-Rating Depression Scale(SDS) | Change from Baseline scores of FDI score at at 3、6、12months after onset.
  The full name of the scale called Zung Self-Rating Depression Scale.The SDS contains 20 questions. Each question is scored on a scale of 1-4 (never, some of the time, relatively often, most of the time). Ten questions involve the assessment of increasing depression levels, and ten questions involve decreasing depression levels.Each items points accumulated as raw scores,the lowest raw score is 20 points, the highest raw score is 80 points. The raw scores multiply by 1.25, taking the integer part as the standard scores.The SAS standard scores were used to define four categories of depression severity: within normal ranger no significant psychopathology (25-49points);presence of mild to moderate depression levels (53-62points); severe depression levels (63-72points); and presence of extreme depression (73-100points).

CONTACTS AND LOCATIONS:
Overall Officials: Bingguo Xu, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No